CLINICAL TRIAL: NCT03130205
Title: Prospective Longitudinal Biomarker Study in Pancreatic Neuroendocrine Tumours
Brief Title: Biomarker Study in Pancreatic Neuroendocrine Tumours
Acronym: PROGRESS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Barbro Eriksson, Professor, Senior Attending, Uppsala University
Other Study IDs: Uppsala University Hospital
Record Dates: First submitted 2017-04-06; First posted 2017-04-26 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Biopsy, Large-Core Needle; Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Core needle Biopsy Phlebotomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Core Needle Biopsy — Core Needle Biopsy is performed from liver metastasis.
Radiation: Computed Tomography — Computed Tomography
Radiation: 18F-FDG-PET — 18F Fluorodeoxyglucose Positron emission tomography
Procedure: Phlebotomy — 3 EDTA tubes drawn from peripheral vein
Genetic: Molecular genetic analysis — Performed on biomaterial from peripheral vein and core needle biopsy

SUMMARY:
The biology of pancreatic neuroendocrine tumors can change during the disease course. This evolution of disease can manifest through increases in tumor proliferation rate, resistance to medical therapy and/or a change in tumor hormone secretion. This study aims to characterize how the biology of pancreatic neuroendocrine tumors change over time, measured by; patient symptoms, biochemistry, contrast enhanced computed tomography, FDG-PET and core needle biopsy with histopathological analysis (Ki67 index and tumor cell differentiation). Uptake on 18F-FDG-PET will be correlated directly to tumor cell proliferation rate. Fraction of patients with spatial heterogeneity in FDG uptake as well as metachronous changes in all collected data will be documented. Biomaterial from whole blood and core needle biopsies will be characterized on the molecular level, and those findings will be integrated to the above specified clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Informed consent
* WHO performance status ≤2
* Progressive disease (as defined by the local investigator) or newly diagnosed disease (defined as prior to medical or oncological intervention except for somatostatin analogue treatment).
* Pathology confirmed diagnosis of pancreatic or duodenal neuroendocrine tumour WHO G1-G3.

  o Exception: In newly diagnosed patients with high suspicion of PNET based on clinical and radiological parameters where tissue sample have not yet been obtained. These patients may be included and subsequently excluded if pathology cannot confirm NET.
* Biopsy procedure not associated with inappropriate risk as determined by the responsible physician.

Exclusion Criteria:

* Patient does not consent
* Permanent risk factors for biopsy

  * Long term treatment with anticoagulant that cannot be temporarily paused without unacceptable risk.
  * Permanent coagulation disorder
* Pregnancy or no contraceptive in fertile women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-resectable metastatic pancreatic neuroendocrine tumors at the Department of Endocrine Oncology, Uppsala, Sweden.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between FDG-PET and tumor biology | Through study completion, an average of 3 years.
  18F-FDG-PET SUVmax correlation to Ki67 index (determined as percentage of tumor cells with positive Ki67 imunohistochemical staining).

CONTACTS AND LOCATIONS:
Overall Officials: Barbro Eriksson, MD PhD, Principal Investigator — Akademiska Sjukhuset, Uppsala
Locations (1):
- Akademiska Sjukhuset, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided